CLINICAL TRIAL: NCT03179644
Title: Study of Variations of Pleural and Esophageal Pressures Under Mechanical Ventilation After Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-08
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Adult patient admitted in the Respiratory Distress and Severe Infections Intensive Care Unit in the postoperative period following a double lung transplant, the objective is to To assess the correlation between the mean pleural pressure and esophageal pressure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bi-pulmonary transplantation (Experimental): Adult patient admitted in the Respiratory Distress and Severe Infections Intensive Care Unit in the postoperative period following a double lung transplant after written informed consent.
  Interventions: Other: Measurement of oesophageal pressure and pleural pressure

INTERVENTIONS:
Other: Measurement of oesophageal pressure and pleural pressure — Measurement of oesophageal pressure by a nasogastric tube with an esophageal balloon (also enabling the patient to be fed) and pleural pressure measurement by means of several pleurocath-type catheters (Prodimed Inc, France) which the thoracic surgeon will have previously Positioned at the end of the surgery without any additional skin intrusion

SUMMARY:
The primary objective of the study is to determine the correlation between mean pleural pressure and oesophageal pressure in the immediate aftermath of bi-pulmonary transplantation.

In this research, oesophageal pressure will be measured by a nasogastric tube with an esophageal balloon (also suitable for feeding the patient) usually installed at the time of transplantation, pleural pressure will be measured by several Pleurocath-type catheters (Prodimed Inc, France) which the thoracic surgeon will have positioned at the end of the surgery without additional skin intrusion.

DETAILED DESCRIPTION:
Pulmonary transplantation is a model of acute lung injury due to ischemia-reperfusion phenomena responsible in 1 in 4 patients for the occurrence of primary graft dysfunction (DPG), which penalizes graft prognosis in the short to medium term. The survival of transplant patients. Furthermore, the post-operative period is a complex period in which multiple hemorrhagic, immunological, infectious, and neuromuscular complications may arise that may require prolonged mechanical ventilation. At present, there are no data on the measurement of pressure in pleural space after pulmonary transplantation. Achieving this measurement would make it possible to adapt the settings of the ventilator to both the acute phase in the case of DPG and to a later phase in case of mechanical weaning. In the case of bi-pulmonary transplantation, before the thorax is closed, each patient benefits from the systematic placement of bilateral anterior and posterior thoracic drains to prevent the formation of fluid effusions (hemothorax, pleurisy) and / or gases (pneumothorax ) Which would impede ventilation and compromise gas exchange. These drains are gradually withdrawn during resuscitation usually after weaning mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

- Adult patient admitted in the Respiratory Distress and Severe Infections Intensive Care Unit in the postoperative period following a double lung transplant after written informed consent.

Exclusion Criteria:

* Age less than 18 years, Pregnancy, breast feeding, adults under guardianship or under safeguard justice, not beneficiaries of a social security scheme, persons deprived of liberty by a judicial or administrative decision , those hospitalized without consent Single lung transplant
* Open chest at the end of transplantation
* high flow pleura-pulmonary fistula (Contraindication to the establishment of a nasogastric tube proven presence of esophageal varices esophageal tumor Surgery of the esophagus of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Oesophageal pressure | 5 days
  The oesophageal pressure will be measured with a nasogastric tube with an esophageal balloon (also enabling the patient to be fed)(6 measurements at the end of inspiration and 6 at the end of expiration).
Pleural pressure | 5 days
  The pleural pressure will be measured using several pleurocath-type catheters (Prodimed Inc, France)(4 inspiratory measures and 4 expiratory measures)

SECONDARY OUTCOMES:
Correlations between the mean pleural pressure and esophageal pressure during the 5 days following a double lung transplant. | 5 days
Comparison between the pleural pressure and esophageal pressure depending on the lung injury, the ventilation mode and the body position (supine and prone position) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital Nord Assistance Publique Hôpitaux de Marseille, Marseille, France